CLINICAL TRIAL: NCT00717353
Title: Genetic Polymorphisms in UGT1A6 and UGT2B7 in Asian Population: Association With Lung Cancer Phenotype
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: NS05/25/04
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Lung cancer

SUMMARY:
Primary

1. To determine the presence and frequency of novel and known UGT1A6 and UGT2B7 polymorphisms in healthy Chinese, Malay and Indian subjects.
2. To determine the presence and frequency of novel and known UGT1A6 and UGT2B7 polymorphisms in Chinese lung cancer patients with squamous cell and adenocarcinoma subtype.
3. To analyze the functional variations in UGT1A6 and UGT2B7 polymorphisms.

Secondary

1 To study the correlation of UGT1A6 and UGT2B7 polymorphisms with lung cancer type.

DETAILED DESCRIPTION:
Germline polymorphisms are inherited genetic variation present in all cells of the body. At molecular level, such variations may affect gene transcription, translation, mRNA stability, protein activity, protein expression (1-3). Mounting evidences have emerged showing that genetic polymorphisms in drug metabolizing genes and DNA repaired genes are major determinants of response to drugs and carcinogens with possible predictive or prognostic value for clinical outcome (4-6). However, only a small number of all polymorphisms discovered have functional significance and it is often difficult to predict this base on nucleotide sequence alone. Genome based studies have generated a wealth of data on genetic polymorphisms far exceeds our knowledge on the function of these variants. Hence, there is an urgent need to characterize the functional and expressional impact of genetic polymorphisms in candidate genes so that appropriate target polymorphisms most likely to affect the phenotype can be selected for larger scale association studies. In this study, we will adopt a novel 2-stage approach to identify and characterize new polymorphisms in the UGT1A6 and 2B7 genes in our Asian population. Data from our initial genotyping work will then be used to optimize the study design of the stage II association study for the generation of hypothesis that lung cancer histology (phenotype) is associated with UGT polymorphisms (genotype). This study will help to advance our understanding in the functional significance and diversity of genetic variants that exist in our population. It may also shed light on the role of UGT in carcinogenesis and will provide vital ground work for future studies of risk assessment, treatment and may allow identification of at risk individual for chemoprevention and adjuvant therapy studies.

ELIGIBILITY:
Inclusion criteria for stage I study

* Subjects >= 18 years old
* Hemoglobin >= 8g/dL, Total white cell counts >3.0 x 103/μl
* ECOG =0

Inclusion criteria for stage II study

* Chinese ethnicity
* Patients >18 years old
* Hemoglobin => 8g/dL, Total white cell counts >3.0 x 103/μl
* Histologically or cytologically confirmed lung cancer for stage II study
* Uncontrolled medical conditions such as diabetes, hypertension and coronary artery disease.

Exclusion criteria

* Histology of small cell lung cancer
* Medical or psychiatric conditions which may impair the patient's ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our laboratory has conducted a pilot study to look at UGT1A expression in both normal and cancer tissue using RT PCR. We have found that in UGT1A6 is the predominant UGT1A enzymes expressed in normal lung and the expression of UGT1A6 enzymes is down regulated in lung cancer (unpublished data). The distribution of UGT1A enzymes in the lung suggests that UGT1A6 may be important in the glucuronidation of inhaled UGT substrates including chemicals from tobacco smoking.
Sampling Method: Probability Sample
Dates: Start 2005-10; Primary Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Desai AA, Innocenti F, Ratain MJ. UGT pharmacogenomics: implications for cancer risk and cancer therapeutics. Pharmacogenetics. 2003 Aug;13(8):517-23. doi: 10.1097/01.fpc.0000054116.14659.e5. PMID 12893990
- [Background] Saeki M, Saito Y, Jinno H, Tanaka-Kagawa T, Ohno A, Ozawa S, Ueno K, Kamakura S, Kamatani N, Komamura K, Kitakaze M, Sawada J. Single nucleotide polymorphisms and haplotype frequencies of UGT2B4 and UGT2B7 in a Japanese population. Drug Metab Dispos. 2004 Sep;32(9):1048-54. PMID 15319348